CLINICAL TRIAL: NCT04052191
Title: Intra-Coronary Administration of MCRcI® (Myo-Cardial Regenerative Cellular Injection) Improves Left Ventricular Function in Patients With Diffuse Coronary Artery Disease
Brief Title: MCRcI® Stem Cell Treatment for Diffuse Coronary Artery Disease
Acronym: MCRcI®
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Honya Medical Inc (Industry)
Collaborators: Chang Gung Memorial Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Single | Purpose: Treatment
Other Study IDs: KCG17121910001
Record Dates: First submitted 2019-08-06; First posted 2019-08-09 (Actual); Last update posted 2024-10-03 (Actual); Status verified 2024-10

CONDITIONS: Coronary Artery Disease
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Intervention Model Description: Dose escalation.
Who Masked: Participant
Masking Description: Participant blind with dose.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Low Dose (Experimental): Low Dose of MCRcI® stem cells.
  Interventions: Biological: MCRcI® stem cells
- Intermediate Dose (Experimental): Intermediate Dose of MCRcI® stem cells.
  Interventions: Biological: MCRcI® stem cells
- High Dose (Experimental): High Dose of MCRcI® stem cells.
  Interventions: Biological: MCRcI® stem cells

INTERVENTIONS:
Biological: MCRcI® stem cells — Intra-Coronary Administration of MCRcI® stem cells
  Other Names: stem cells

SUMMARY:
Safety evaluation of Intra-Coronary Administration of MCRcI® stem cells in Patients with Diffuse Coronary Artery Disease.

ELIGIBILITY:
Inclusion Criteria:

* Patients with Diffuse Coronary Artery Disease
* Age 20~80
* Participants have received proper medication
* Canadian Cardiovascular Society class II- IV Angina.

Exclusion Criteria:

* Age <20 or >80
* Pregnant or breast feeding
* Positive adventitious infection (such as HIV, hepatitis )
* History of Myocardial Infarction within past 3 months
* Severe aortic or mitral valve narrowing
* Short of breath unable to receive PCI examination or treatment
* Malignant tumor
* Hematopoietic dysplasia
* Severe organ disease with less than 1 year of life expectancy
* Chronic kidney disease with CCr<20ml/min
* Kiney disease on renal dialysis.

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-12-01 (Estimated); Primary Completion 2026-01-01 (Estimated); Study Completion 2026-12-01 (Estimated)

PRIMARY OUTCOMES:
Incidence of Treatment Emergent Adverse Events | 6 months
  Number of adverse events

SECONDARY OUTCOMES:
Left ventricle stroke volume | 12 months
  Echocardiogram assessment on left ventricle stroke volume (volume of blood pumped from the left ventricle per beat (ml).
End diastolic volume | 12 months
  Echocardiogram assessment on volume of blood in the left ventricle at the end of diastolic filling (ml)
Left ventricular ejection fraction (LVEF) | 12 months
  Calculated by dividing the volume of blood pumped from the left ventricle per beat (stroke volume) by the volume of blood collected in the left ventricle at the end of diastolic filling (end-diastolic volume).
Severity of angina symptom using Canadian Cardiovascular Society grading. | 12 months
  Canadian Cardiovascular Society grading of angina pectoris is a classification system used to grade the severity of exertional angina. Scale ranges 0 ~ IV (most sever), with 0 Asymptomatic Angina, I Angina only with strenuous exertion, II Angina with moderate exertion, III Angina with mild exertion and IV Angina at rest.

CONTACTS AND LOCATIONS:
Overall Officials: Fang Y Lee, MD, Principal Investigator — Chang Gung Memorial Hospital
Locations (1):
- HONYA Medical Inc, Tainan, Taiwan

IPD SHARING:
Plan to Share IPD: No